CLINICAL TRIAL: NCT00309088
Title: FK506 Phase 3 Study: a Double Blind Placebo Controlled Study for Steroid Non-Resistant Myasthenia Gravis Patients
Brief Title: FK506 Phase 3 Study: a Study for Steroid Non-resistant Myasthenia Gravis (MG) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F506-CL-0601
Record Dates: First submitted 2006-03-29; First posted 2006-03-31 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Myasthenia Gravis
Keywords: Tacrolimus; Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tacrolimus
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tacrolimus — oral
  Other Names: Prograf; FK506
  Arms: 1
Drug: placebo — oral
  Arms: 2

SUMMARY:
The purpose of the study is to investigate the efficacy and safety for steroid non-resistant MG patients in a double blind, placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as myasthenia gravis
* Those whose MG symptoms are well-controlled by the treatment with prednisone
* Steroid non-refractory Myasthenia Gravis: ≧20mg and ≦40mg / alternate day of steroid dose required to maintain

Exclusion Criteria:

* Those who have thymoma or the history of thymoma (Masaoka stage III or IV)
* Patients who received steroid pulse therapy, plasma exchange therapy, globulin therapy or radiation therapy within 12 weeks prior to the initiation of test drug
* Patients who started the immunosuppressant therapy or increased the dose of immunosuppressant within 12 weeks prior to the initiation of test drug.
* Patients who had undergone thymectomy within 24 weeks prior to the initiation of test drug.
* Pancreatitis or diabetes
* Serum creatinine≦1.5mg/dL

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2006-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Mean dose of steroid to maintain minimal manifestation(MM)[The dose of steroid should be decreased by the rate of 5mg/alternate day/ 4 weeks after the initiation of tacrolimus or placebo treatment as far as the MM state should be maintained.] | 6 Months

SECONDARY OUTCOMES:
Total amount of steroid therapy (mg) | 6 Months
QMG score;MG-ADL | 6 Months
Success rate of achievement to the targeted steroid dose | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (9):
- Japan (9):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Hokuriku Region
  - Kansai Region
  - Kanto Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

REFERENCES:
- [Derived] Yoshikawa H, Kiuchi T, Saida T, Takamori M. Randomised, double-blind, placebo-controlled study of tacrolimus in myasthenia gravis. J Neurol Neurosurg Psychiatry. 2011 Sep;82(9):970-7. doi: 10.1136/jnnp-2011-300148. Epub 2011 Jul 22. PMID 21784757